CLINICAL TRIAL: NCT01705314
Title: Effect of Vitamin D3 Supplementation to Reduce Respiratory Infections in Children and Adolescents in Vietnam: A Blinded, Placebo-controlled Randomized Controlled Trial
Brief Title: A Randomized Trial of Vitamin D to Reduce Respiratory Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: VitD2012
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Respiratory Infection
Keywords: human influenza children
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D supplements (Experimental): children and adolescents that are randomized to the intervention will receive 7 mls of D-drops (14,000U/week of vitamin D) for eight months
  Interventions: Dietary Supplement: vitamin D supplements
- vitamin D placebo (Placebo Comparator): children and adolescents that are randomized to placebo will receive 7 mls of placebo drops for eight months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamin D supplements — Participants will receive 7mls of D-drops (14,000U/week of vitamin D)
  Arms: vitamin D supplements
Dietary Supplement: placebo — 7mls of placebo drops per week for 8 months.
  Arms: vitamin D placebo

SUMMARY:
The goal of this study is to assess the effectiveness of vitamin D in reducing laboratory-confirmed influenza and in reducing non-influenza viral respiratory tract infections. A cohort of children between the ages of 3 and 17 years from the Thanh Ha Commune, Thanh Liem District, Ha Nam Province, Vietnam will be randomized to either weekly vitamin D supplements or placebo. Participants who develop acute respiratory infection over a 12-month period, will be tested for influenza, the co-primary outcome, and other respiratory viruses, the other co-primary outcome, by RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 3 and 17
* Residing in Thanh Liem District, Ha Nam Province, Vietnam

Exclusion Criteria:

* Born prematurely at less than 32 weeks gestation
* Any chronic illness (except asthma)
* Currently using medication known to interfere with vitamin D metabolism
* Children with a sibling participating in the study

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1300 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed non-influenza infection | 12 months
Laboratory-confirmed influenza infection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, Principal Investigator — McMaster University, Hamilton, ON, Canada
Locations (1):
- National Institute of Hygiene and Epidemiology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No